Cover Page for IRB Approval Document
Official Study Title: What makes people better at retrieving proper names?
NCT05550779

Document Date: 7/10/2024



## University of Colorado Colorado Springs (UCCS) Consent to be a Research Subject

Title: What makes people better at retrieving names of famous people?

Principal Investigator: Hannah Levitt

Funding Source: National Institutes of Health

Key Information You are being asked to choose whether or not you would like to participate in a research study. This study is being conducted to learn more about how various personal and situational characteristics are related to the ability to produce names of famous people in response to photographs. You will listen to an audio clip, then see photographs of famous people and try to come up with the name that fits each one. You will also complete some surveys and other measures. Participation will take approximately 60–75 minutes. There are minimal risks involved in this study, but you may feel frustrated by the difficulty of the name retrieval task, or you might become bored with the audio clip or surveys. Collected data will be stored by an identification code, not your name. You will not directly benefit from this study, but it will give researchers a better understanding of how individuals' personality and cognitive traits and setting in which naming occurs correspond with their ability to produce names.

<u>Introduction</u> You are being asked to be in a research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) to be in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study.

Before making your decision:

- Please carefully read this form or have it read to you.
- Please ask questions about anything that is not clear.

Feel free to take your time thinking about whether you would like to participate. By agreeing to be in the study you will not give up any legal rights. You may want to print a copy of the consent form for your records.

<u>Study Overview</u> This study is being conducted to learn more about how various personal and situational factors relate to the ability to produce names that fit photographs. Results will be presented as group averages, not as individual responses. Findings may be published in journal articles and presented at conferences.

<u>Procedures</u> You are being asked to be in this research study because you are 18–35 or 60–80 years of age, a native, fluent speaker of American English, and have lived in the United States for at least 5 years. If you choose to participate, you will engage in a videoconference call with a researcher and complete some surveys on Qualtrics. You will first listen to a

brief audio clip, following which you will be asked to provide names that fit the photographs. We will video record the name retrieval task for later scoring verification. People over the age of 60 will complete one additional set of cognitive questions at the end of the study. The entire procedure will take approximately 60-75 minutes to complete.

Other people in this study: 120 people will participate in this study.

<u>Risks and Discomforts</u> There is minimal risk involved in this study. You might feel frustrated by the name retrieval task, or you might become bored while doing the exercise with the audio clip or while completing the surveys. You may stop participating in the study at any time without any negative consequences.

<u>Benefits</u> You will not directly benefit from this study, but it will give researchers a better understanding of how individuals' personal traits and situational factors relate to the ability to produce names of famous faces.

<u>Compensation</u> UCCS student participants are compensated with 2.5 SONA system credits. Non-student participants are compensated with a \$15 electronic gift certificate.

Confidentiality None of your data will have your name attached to it, nor will the video recording. Participant information will be kept separately from data, in a secure location. Participant information and data will be stored only by a meaningless participant identification code. Only Hannah Levitt, her faculty advisor (Dr. Lori James), and her research assistants will have access to raw or coded data. All electronic data files will be kept on password-protected computers.

Certain offices and people other than the researchers may have access to study records. Government agencies and UCCS employees overseeing proper study conduct may look at your study records. These offices include the UCCS Institutional Review Board, and the UCCS Office of Sponsored Programs and Research Integrity. UCCS will keep any research records confidential to the extent allowed by law. A participant identification code rather than your name will be used on study records wherever possible. Study records may be subject to disclosure pursuant to a court order, subpoena, law or regulation.

Your de-identified data collected during this study could be used for future research studies without additional consent. Also, your de-identified data may be made available to the scientific community in an online format as required by sponsors or publishers.

## Voluntary Participation and Withdrawal from the Study

Taking part in this study is voluntary. You have the right to leave the study at any time without penalty. You may refuse to answer any questions that

you do not wish to answer. If you withdraw from the study, you may request that your data not be used by contacting the Principal Investigator listed above and below. If you are a UCCS student, there are alternative options to earn credit other than participating in this study. Contact your course instructor if you would like to learn about alternatives for receiving extra credit.

## Contact Information

Contact (PI's info): Contact (PI's info): Hannah Levitt at hlevitt@uccs.edu

- if you have any questions about this study or your part in it,
- if you have questions, concerns or complaints about the research, or
- if you would like information about the survey results when they are prepared.

Contact the Research Integrity Compliance Program Director at 719–2553903 or via email at irb@uccs.edu:

- · if you have questions about your rights as a research participant, or
- if you have questions, concerns or complaints about the research.

<u>Electronic Consent</u> Please print a copy of this consent form for your records, if you so desire.

I have read and understand the above consent form, I certify that I am 18 years old or older and, by verballing consenting to the study and having the researcher click the "Agree" and submit buttons, I indicate my willingness to voluntarily take part in the study.